CLINICAL TRIAL: NCT04570943
Title: Phase II Study to Assess the Interest of a Sequential Treatment With Gemcitabine/Nab-paclitaxel (GEMBRAX) and Then FOLFIRINOX Followed by Stereotactic Magnetic Resonance-guided Adaptive Radiotherapy in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Sequential Treatment With GEMBRAX and Then FOLFIRINOX Followed by Stereotactic MRI-guided Radiotherapy in Patients With Locally Advanced Pancreatic Cancer
Acronym: GABRINOX-ART
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROICM 2020-04 GAB
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-04

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma
Keywords: Pancreatic; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gabrinox followed by stereotactic radiotherapy (Experimental): Gembrax:
  Albumin-bound paclitaxel followed by Gemcitabine Day 1,8,15 followed by 2 weeks of rest
  Folfirinox:
  Oxaliplatin, irinotecan, leucovorin, 5FU bolus and continuous
  Interventions: Combination Product: Gabrinox; Radiation: MRI-GUIDED STEREOTACTIC RADIOTHERAPY

INTERVENTIONS:
Combination Product: Gabrinox — Regimen: GEMBRAX
  Other Names:
  Albumin bound paclitaxel 125 mg/m² + Gemcitabine 1000 mg/m²
  Regimen: FOLFIRINOX
  Other Names:
  Oxaliplatin 85 mg/m² + Leucovorin 200 mg/m² + Irinotecan 180 mg/m² + 5FU bolus 400mg/m² + 5FU continuous 2400 mg/m²
  Gembrax + Folfirinox = GABRINOX
Radiation: MRI-GUIDED STEREOTACTIC RADIOTHERAPY — Radiotherapy will start between 5 and 6 weeks after the last injection of chemotherapy (FOLFIRINOX regimen) in non-progressive patients after Gabrinox.
  Stereotactic adaptive radiotherapy in five fractions: prescription dose in five fractions of 10 Gy/day on consecutive days. At least two sessions/week should be performed. An interval of at least 18 hours between fractions is recommended.

SUMMARY:
The aim of this study is to demonstrate the efficacy of intensified and sequential chemotherapy (Gabrinox) comprising Gembrax regimen (Gemcitabine-Abraxane) followed by the Folfirinox regimen (5FU, Oxaliplatin and Irinotecan) in patients with locally advanced pancreatic adenocarcinoma.

The study will also demonstrate the feasibility of combining this intensified chemotherapy with MRI-guided stereotactic radiotherapy in non-progressive patients after the chemotherapy by Gabrinox regimen.

DETAILED DESCRIPTION:
Pancreatic cancer was the third cause of death by cancer worldwide in 2016, surpassing breast cancer. It is estimated that in 2030, pancreatic cancer will become the second cause of death by cancer after lung cancer.

Its prognosis is very poor, with an overall survival (OS) at 5 years, all stages included, of 5.5%. According to the French cancer registry network (FRANCIM), its incidence has more than doubled in men and women between 1990 and 2018. The world standardized incidence rates for men and women were 5.2% and 2.7% in 1990 and 11% and 7% in 2018, respectively. This means a yearly annual increase of 2.7 for men and of 3.8 for women. The often late diagnosis, in 50% of cases at stage 4, and the limited treatment options explain the very low survival rate at 5 years.

Currently, only surgery associated with adjuvant chemotherapy for 6 months allows doubling this survival rate. However, this situation concerns only 20% of cases. Indeed, 50% of pancreatic cancers are discovered at stage 4, and in 30% of patients cancer is detected when not resectable and non-metastatic (i.e. borderline resectable or locally advanced). To make an unresectable cancer resectable is one of the therapeutic strategies under development. However, treatment of locally advanced pancreatic cancer (LAPC) is not standardized. Chemotherapy is a used strategy, but 30% of cases will progress to metastatic disease. Therefore, the need in LAPC to control not only the local disease but also micro-metastases has led to the development of combined strategies with chemotherapy and optimal radiotherapy.

For LAPC, chemotherapy is based on two drug combinations that are classically used for the first-line treatment of metastatic disease: FOLFIRINOX (FFX) (association of 5FU, Oxaliplatin and Irinotecan) and GEMBRAX (GA) (association of gemcitabine and nab-paclitaxel). Their association has been validated by phase 3 studies showing that compared with gemcitabine alone, they allow increasing the response rate by three times (30%), and almost doubling the median survival and progression-free survival, but with higher grade 3 hematologic and neurological toxicities.

FFX and GA have been assessed also in LAPC. Retrospective studies confirmed the high response rate, 30 to 80% according to the study, and a median survival of 9 to 30 months. Recently, two phase 2 studies, evaluated GA alone and GA followed by FFX, respectively, for LAPC, and confirmed the efficacy, with a response rate of 30% and a secondary resection rate of 15% and 30.6%, respectively. Moreover, in patients who underwent tumour resection after treatment, survival was longer than in those not operated (27.4 vs 14.2 months; Hazard Ratio (HZ) = 0.45; p = 0.0035). Overall Survival (OS) (n= 165 patients) was 17.2 months.

GABRINOX is a sequential treatment with GA and then FFX with the aim of limiting chemoresistance, decreasing toxicities and improving dose intensity.

The feasibility and tolerance of this approach as first-line treatment of metastatic disease were validated in a phase 1 study, and its efficacy in a phase 2 study in which the primary objective was reached: objective response rate of 64.9%, disease control rate of 84.2%, progression-free survival (PFS) of 10.5 months, and Overall Survival (OS) of 15.1 months. Its tolerance profile is favorable with lower percentages of patients with neutropenia (34.5%), febrile neutropenia (3.5%), and neurotoxicity (5.2%).

The role of chemo-radiotherapy for LAPC remains controversial. Many old studies showed the interest of this technique for the local and global control in patients with pancreatic cancer.

However, a phase 3 study compared the efficacy of chemo-radiotherapy versus chemotherapy alone in patients without disease progression after chemotherapy with a regimen that is currently considered not optimal (i.e. gemcitabine with/without erlotinib). Although OS (the main endpoint) did not improve in the chemo-radiotherapy arm compared with the chemotherapy arm, PFS was significantly increased in the chemo-radiotherapy arm with a longer period without treatment (6.1 vs 3.7 months, P = 0.02) and a lower percentage of patients with locoregional progression (32% vs 46%, P =0.03). This confirms that radiotherapy is an effective treatment in pancreatic adenocarcinoma, but that the current delivery modalities do not allow significantly improving the patient prognosis. Indeed, the study used 3D conformal radiotherapy with conventional doses and classical fractioning. Retrospective and phase 1 and 2 studies that used more optimized techniques and higher doses reported better local disease control, but without an important impact on survival. Moreover, some studies suggest significant toxicity, particularly in gastrointestinal organs. Intensity-modulated radiotherapy and integrated boost radiotherapy showed promising local control and survival results. This suggests an avenue for technological improvement and dose augmentation to improve patient prognosis.

Stereotactic magnetic resonance-guided adaptive radiotherapy is a new modality for dose delivery that exploits Magnetic Resonance Imaging (MRI)-guided linear accelerators to better target the treatment volume, while optimizing the protection of organs at risk. The tumour localization in the pancreas seems to be particularly suitable for the utilization of MRI-guided linear accelerators because the radiotherapy doses are limited in function of the gastrointestinal organ tolerance: duodenum, stomach, small intestine, colon. Recently, the results of a retrospective, multicentre study on irradiation of patients with LAPC using Magnetic Resonance Imaging (MRIdian® Linac™; Viewray. The study shows that survival was improved in patients who received an augmented irradiation dose. Specifically, the 2-year OS rate was 49% for patients who received a dose higher than 70 Gy and 30% for patients who received a lower equivalent dose. The study did not report significant toxicity in patients who received high-dose radiotherapy according to the optimized modalities with daily dosimetric adjustment and target monitoring at each radiotherapy session. These data suggest that dose intensification and the stereotactic magnetic resonance-guided adaptive radiotherapy technique improve radiotherapy results; however, prospective studies are needed to confirm these data.

Therefore, the phase 2 study GABRINOX-ART in which an intensified chemotherapy regimen (GABRINOX i.e GA followed by FFX) is followed by optimized adjusted radiotherapy (stereotactic magnetic resonance-guided adaptive radiotherapy) seems to be an interesting strategy to evaluate in locally advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged from 18 to 75 years at the date of signature of the consent form
2. Histologically or cytologically proven pancreatic adenocarcinoma
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
4. Non-resectable tumour according to the National Comprehensive Cancer Network (NCCN) 1.2015 recommendations after external review of imaging data by multidisciplinary experts.
5. Non-metastatic cancer confirmed by thorax-abdomen-pelvis computerized tomography (CT) scan and liver MRI
6. SMART feasibility confirmed by centralized review
7. Uracilemia < 16 ng/ml
8. Hematological assessment within 14 days before inclusion, defined by:

   * Neutrophils ≥ 2 000/mm3 (2 × 109/L);
   * Platelets ≥ 100 000/mm3 (100 × 109/L);
   * Hemoglobin ≥ 9 g/dl
9. Liver function (within 14 days before inclusion) defined by:

   * ASpartate Transaminase (AST) and ALanine Transaminase (ALT) ≤ 2.5 x Upper Limit of Normal (ULN);
   * Total bilirubin ≤ 1.5 x ULN. Patients with a metallic biliary prosthesis due to biliary obstruction caused by the cancer may be included, if: a CT scan with injection of contrast medium and thin pancreas sections was performed before placing the biliary prosthesis, the bilirubin level after prosthesis fitting decreased to ≤20 mg/L (≤34 μmol/L), and in the absence of cholangitis.
10. Creatininaemia within the reference limits, or calculated clearance ≥50 ml/min for patients with a serum creatinine value above or below the reference values (clearance calculated using the Chronic Kidney Disease EPIdemiology collaboration (CKDEPI formula).
11. Serum calcium AND magnesium AND potassium ≥ Lower Limit Normal (LLN and ≤ 1.2 x Upper Limit Normal (ULN)
12. Cancer Antigen (CA 19.9) <500 IU/mL (without cholestasis). Patients with CA 19.9 between 500 IU/mL and 1000 IU/mL can be included if the Positron Emission Tomography (PET) scan and peritoneal MRI (optional) do not detect any distant fixation, indicative of metastasis. Patients with CA 19.9 ≥ 1000 IU/mL cannot be included.
13. Sexually active patients must use a contraceptive method considered adequate and suitable by the investigator during the entire period of administration of the study treatment and up to 6 months after the treatment end, for female and male patients.
14. Signature of the consent form before any study-specific procedure.
15. Covered by the French health insurance.

Exclusion Criteria:

1. Any previous treatment for pancreatic cancer (e.g. chemotherapy, radiotherapy, surgery, targeted therapy, experimental therapy)
2. Gilbert's syndrome or homozygous Uridine DiPhosphate Glucuronosyl Transferase 1 A1 (UGT1A1 * 28)
3. Other concomitant cancer or history of cancer, except for treated in situ cancer of the cervix , basal cell or squamous cell carcinoma, superficial bladder tumour (Ta, Tis, and T1), or good-prognosis tumour cured without chemotherapy and without signs of disease in the 3 years before inclusion
4. Prior radiotherapy likely to overlap with the planned study radiotherapy area (e.g. previous abdominal irradiation).
5. Patients with high cardiovascular risk, including, but not limited to, coronary stent or myocardial infarction in the past 6 months.
6. Peripheral neuropathy ≥ grade 2
7. ECG with QTcorrected (QTc) interval longer than 450 ms for men and longer than 470 ms for women
8. Contraindication to MRI and MRI-guided radiotherapy
9. History of chronic inflammatory disease of the colon or rectum
10. Any other concomitant and not controlled serious illness or disturbance that may interfere with the patient's participation in the study and safety during the study (e.g. severe liver, kidney, lung, metabolic, or psychiatric disorder)
11. Intolerance or allergy to one of the study drugs (gemcitabine, Nab-paclitaxel, oxaliplatin, irinotecan, 5-FU) or to one of their excipients (e.g. fructose) listed in the Contraindications or Warnings sections and Special precautions of the Summary of Product Characteristics (SmPC) or prescription information
12. Legal incapacity (patient under guardianship or wardship)
13. Pregnant or breastfeeding woman. Fertile women must have a negative pregnancy test (serum β-hCG) performed 72 hours before inclusion
14. Patient using vitamin K antagonists (Coumadin…) (possible modification of the treatment before inclusion)
15. Active and uncontrolled bacterial or fungal infection that requires systemic treatment.
16. Know active HIV infection
17. History of peripheral arterial disease (e.g. lameness, Buerger's disease).
18. Patient who received a attenuated live vaccine in the 10 days before inclusion
19. Patient with history of pulmonary fibrosis or interstitial pneumonia.
20. Inability to attend the follow-up visits due to geographic, social or mental reasons.
21. Participation in another clinical study with a research product during the last 30 days before inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Rate of non-progression at 4 months | 4 months
  (Sequence 1 success = chemotherapy) according to the RECIST v1.1 criteria
Acute gastrointestinal non-toxicity rate | 90 days
  Absence of toxicity of grade ≥3 related to radiotherapy within 90 days, evaluated using the NCI-CTCAE v5.0 classification (sequence 2 success = radiotherapy)

SECONDARY OUTCOMES:
Assessment of adverse events due to chemotherapy by using the NCI-CTCAE version 5.0 scale | 36 months
  Adverse events of chemotherapy evaluated using the NCI-CTCAE v5.0 classification
Assessment of adverse events due to radiotherapy by using the NCI-CTCAE version 5.0 | 36 months
  Adverse events of radiotherapy evaluated using the NCI-CTCAE v5.0 classification
Collection of dosimetric results regarding dose/volume from the planned dosimetry, such as coverage of the planning targeted volume (PTV) by the prescription dose in the accumulated dose | An average of 9 months after the beginning of treatment (chemotherapy then radiotherapy)
  End of radiotherapy
Collection of dosimetric results regarding dose/volume from the planned dosimetry, such as dose received by the gross total volume | An average of 9 months after the beginning of treatment (chemotherapy then radiotherapy)
  End of radiotherapy
Collection and Summation of the dosimetric results in terms of dose/volume for the adaptive radiotherapy sessions and comparison with the predicted dosimetry | An average of 9 months after the beginning of treatment (chemotherapy then radiotherapy)
  End of radiotherapy
Correlation of the dose received by organs at risk (duodenum, small intestine, stomach, colon) with the appearance of gastrointestinal toxicities | An average of 9 months after the beginning of treatment (chemotherapy then radiotherapy)
  End of radiotherapy
Correlation of planning target volume (PTV) coverage and dose received by the gross tumor volume (GTV) with progression free survival | An average of 9 months after the beginning of treatment (chemotherapy then radiotherapy)
  End of radiotherapy
Correlation of planning target volume (PTV) coverage and dose received by the gross tumor volume (GTV) with overall survival | An average of 9 months after the beginning of treatment (chemotherapy then radiotherapy)
  End of radiotherapy
Progression-free Survival (PFS) of the radiotherapy | Through study completion, an average of 68 months
  Between the radiotherapy start date and the date of the first documented progression or the date of death from any cause
Overall Survival (OS) of the radiotherapy | Through study completion, an average of 72 months
  Interval between the radiotherapy start date and the date of death from any cause
Local disease control of the radiotherapy | Through study completion, an average of 68 months
  Interval between the radiotherapy start date and the date of local progression of the disease
Progression-free Survival (PFS) of the whole treatement | Through study completion, an average of 72 months
  Between the date of inclusion and the date of the first documented progression or the date of death from any cause
Overall Survival (OS) of the whole treatement | Through study completion, an average of 72 months
  Interval between the date of inclusion and the date of death from any cause
Assessment of adverse events due to the whole treatement | Through study completion, an average of 36 months
  Assessment of adverse events by using the NCI-CTCAE version 5.0 scale from inclusion of first patient until the end of treatment
Resection rate | From the end of radiotherapy (3 months) through 6 months post-radiotherapy
  Percentage of patients who undergo tumour surgery up to 6 months post-radiotherapy
Healthy margin resection rate (R0) | From the end of radiotherapy (3 months) through 6 months post-radiotherapy
Histological response rate | From the end of radiotherapy (3 months) through 6 months post-radiotherapy
  Histological response rate according to the College of American Pathologists grading system.
Prognostic impact of CA 19-9 changes on survival | Through study completion, an average of 36 months
Quality of life by using the quality of life questionnaire score (QLQ-C30) | Through study completion, an average of 60 months
  The EORTC QLQ-C30 uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
  The EORTC QLQ-C30 uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.
Quality of life by using the quality of life questionnaire score (QLQ-PAN26) | Through study completion, an average of 60 months
  The QLQ-PAN26 uses for the question 31 to 56 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much").

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Portalès, MD, Study Chair — Institut de Cancérologie de Montpellier (ICM)
Locations (9):
- France (9):
  - Institut Paoli Calmettes, Marseille, Bouches-du-Rhône
  - CHU Carémeau, Nîmes, Gard
  - CHU Saint-Eloi, Montpellier, Herault
  - Institut régional du Cancer de Montpellier, Montpellier, Hérault
  - Hôpital Beaujon, Clichy
  - Centre Georges-François Leclerc, Dijon
  - Hôpital Pitié Salpétriêre, Paris
  - Centre Eugène Marquis, Rennes
  - Hopital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
All data will be available after publication of the results in peer-reviewed revues, and in national and international meetings. It includes all de-identified participants' data, the study protocol, the statistical analysis plan and the clinical study report. The corresponding author will provide data and datasets generated and/or analyzed during the study upon reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to study data upon written detailed request sent to ICM, from 6 months until 5 years after publication of summary data.
Access Criteria: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from ICM for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Ferlay J, Partensky C, Bray F. More deaths from pancreatic cancer than breast cancer in the EU by 2017. Acta Oncol. 2016 Sep-Oct;55(9-10):1158-1160. doi: 10.1080/0284186X.2016.1197419. Epub 2016 Aug 23. PMID 27551890
- [Background] Conroy T, Hammel P, Hebbar M, Ben Abdelghani M, Wei AC, Raoul JL, Chone L, Francois E, Artru P, Biagi JJ, Lecomte T, Assenat E, Faroux R, Ychou M, Volet J, Sauvanet A, Breysacher G, Di Fiore F, Cripps C, Kavan P, Texereau P, Bouhier-Leporrier K, Khemissa-Akouz F, Legoux JL, Juzyna B, Gourgou S, O'Callaghan CJ, Jouffroy-Zeller C, Rat P, Malka D, Castan F, Bachet JB; Canadian Cancer Trials Group and the Unicancer-GI-PRODIGE Group. FOLFIRINOX or Gemcitabine as Adjuvant Therapy for Pancreatic Cancer. N Engl J Med. 2018 Dec 20;379(25):2395-2406. doi: 10.1056/NEJMoa1809775. PMID 30575490
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Suker M, Beumer BR, Sadot E, Marthey L, Faris JE, Mellon EA, El-Rayes BF, Wang-Gillam A, Lacy J, Hosein PJ, Moorcraft SY, Conroy T, Hohla F, Allen P, Taieb J, Hong TS, Shridhar R, Chau I, van Eijck CH, Koerkamp BG. FOLFIRINOX for locally advanced pancreatic cancer: a systematic review and patient-level meta-analysis. Lancet Oncol. 2016 Jun;17(6):801-810. doi: 10.1016/S1470-2045(16)00172-8. Epub 2016 May 6. PMID 27160474
- [Background] Philip PA, Lacy J, Portales F, Sobrero A, Pazo-Cid R, Manzano Mozo JL, Kim EJ, Dowden S, Zakari A, Borg C, Terrebonne E, Rivera F, Sastre J, Bathini V, Lopez-Trabada D, Asselah J, Saif MW, Shiansong Li J, Ong TJ, Nydam T, Hammel P. Nab-paclitaxel plus gemcitabine in patients with locally advanced pancreatic cancer (LAPACT): a multicentre, open-label phase 2 study. Lancet Gastroenterol Hepatol. 2020 Mar;5(3):285-294. doi: 10.1016/S2468-1253(19)30327-9. Epub 2020 Jan 14. PMID 31953079
- [Background] Kim YJ, Lee WJ, Woo SM, Kim TH, Han SS, Kim BH, Moon SH, Kim SS, Koh YH, Park SJ, Kim JY, Kim DY, Park JW. Comparison of capecitabine and 5-fluorouracil in chemoradiotherapy for locally advanced pancreatic cancer. Radiat Oncol. 2013 Jul 3;8:160. doi: 10.1186/1748-717X-8-160. PMID 23822606
- [Background] Huang J, Robertson JM, Margolis J, Balaraman S, Gustafson G, Khilanani P, Nadeau L, Jury R, McIntosh B. Long-term results of full-dose gemcitabine with radiation therapy compared to 5-fluorouracil with radiation therapy for locally advanced pancreas cancer. Radiother Oncol. 2011 May;99(2):114-9. doi: 10.1016/j.radonc.2011.05.038. Epub 2011 May 27. PMID 21621866
- [Background] Mukherjee S, Hurt CN, Bridgewater J, Falk S, Cummins S, Wasan H, Crosby T, Jephcott C, Roy R, Radhakrishna G, McDonald A, Ray R, Joseph G, Staffurth J, Abrams RA, Griffiths G, Maughan T. Gemcitabine-based or capecitabine-based chemoradiotherapy for locally advanced pancreatic cancer (SCALOP): a multicentre, randomised, phase 2 trial. Lancet Oncol. 2013 Apr;14(4):317-26. doi: 10.1016/S1470-2045(13)70021-4. Epub 2013 Mar 6. PMID 23474363
- [Background] Yang YF, Cao XH, Bao CE, Wan X. Concurrent radiotherapy with oral fluoropyrimidine versus gemcitabine in locally advanced pancreatic cancer: a systematic review and meta-analysis. Onco Targets Ther. 2015 Nov 9;8:3315-22. doi: 10.2147/OTT.S91292. eCollection 2015. PMID 26635481
- [Background] Hammel P, Huguet F, van Laethem JL, Goldstein D, Glimelius B, Artru P, Borbath I, Bouche O, Shannon J, Andre T, Mineur L, Chibaudel B, Bonnetain F, Louvet C; LAP07 Trial Group. Effect of Chemoradiotherapy vs Chemotherapy on Survival in Patients With Locally Advanced Pancreatic Cancer Controlled After 4 Months of Gemcitabine With or Without Erlotinib: The LAP07 Randomized Clinical Trial. JAMA. 2016 May 3;315(17):1844-53. doi: 10.1001/jama.2016.4324. PMID 27139057
- [Background] Petrelli F, Comito T, Ghidini A, Torri V, Scorsetti M, Barni S. Stereotactic Body Radiation Therapy for Locally Advanced Pancreatic Cancer: A Systematic Review and Pooled Analysis of 19 Trials. Int J Radiat Oncol Biol Phys. 2017 Feb 1;97(2):313-322. doi: 10.1016/j.ijrobp.2016.10.030. Epub 2016 Oct 24. PMID 28068239
- [Background] Reyngold M, Parikh P, Crane CH. Ablative radiation therapy for locally advanced pancreatic cancer: techniques and results. Radiat Oncol. 2019 Jun 6;14(1):95. doi: 10.1186/s13014-019-1309-x. PMID 31171025
- [Background] Crane CH, O'Reilly EM. Ablative Radiotherapy Doses for Locally Advanced: Pancreatic Cancer (LAPC). Cancer J. 2017 Nov/Dec;23(6):350-354. doi: 10.1097/PPO.0000000000000292. PMID 29189331
- [Background] Acharya S, Fischer-Valuck BW, Kashani R, Parikh P, Yang D, Zhao T, Green O, Wooten O, Li HH, Hu Y, Rodriguez V, Olsen L, Robinson C, Michalski J, Mutic S, Olsen J. Online Magnetic Resonance Image Guided Adaptive Radiation Therapy: First Clinical Applications. Int J Radiat Oncol Biol Phys. 2016 Feb 1;94(2):394-403. doi: 10.1016/j.ijrobp.2015.10.015. Epub 2015 Oct 17. PMID 26678659
- [Background] Fischer-Valuck BW, Henke L, Green O, Kashani R, Acharya S, Bradley JD, Robinson CG, Thomas M, Zoberi I, Thorstad W, Gay H, Huang J, Roach M, Rodriguez V, Santanam L, Li H, Li H, Contreras J, Mazur T, Hallahan D, Olsen JR, Parikh P, Mutic S, Michalski J. Two-and-a-half-year clinical experience with the world's first magnetic resonance image guided radiation therapy system. Adv Radiat Oncol. 2017 Jun 1;2(3):485-493. doi: 10.1016/j.adro.2017.05.006. eCollection 2017 Jul-Sep. PMID 29114617
- [Background] Henke LE, Contreras JA, Green OL, Cai B, Kim H, Roach MC, Olsen JR, Fischer-Valuck B, Mullen DF, Kashani R, Thomas MA, Huang J, Zoberi I, Yang D, Rodriguez V, Bradley JD, Robinson CG, Parikh P, Mutic S, Michalski J. Magnetic Resonance Image-Guided Radiotherapy (MRIgRT): A 4.5-Year Clinical Experience. Clin Oncol (R Coll Radiol). 2018 Nov;30(11):720-727. doi: 10.1016/j.clon.2018.08.010. Epub 2018 Sep 7. PMID 30197095
- [Background] Henke L, Kashani R, Robinson C, Curcuru A, DeWees T, Bradley J, Green O, Michalski J, Mutic S, Parikh P, Olsen J. Phase I trial of stereotactic MR-guided online adaptive radiation therapy (SMART) for the treatment of oligometastatic or unresectable primary malignancies of the abdomen. Radiother Oncol. 2018 Mar;126(3):519-526. doi: 10.1016/j.radonc.2017.11.032. Epub 2017 Dec 23. PMID 29277446
- [Background] Boldrini L, Cusumano D, Cellini F, Azario L, Mattiucci GC, Valentini V. Online adaptive magnetic resonance guided radiotherapy for pancreatic cancer: state of the art, pearls and pitfalls. Radiat Oncol. 2019 Apr 29;14(1):71. doi: 10.1186/s13014-019-1275-3. PMID 31036034
- [Background] Bohoudi O, Bruynzeel AME, Meijerink MR, Senan S, Slotman BJ, Palacios MA, Lagerwaard FJ. Identification of patients with locally advanced pancreatic cancer benefitting from plan adaptation in MR-guided radiation therapy. Radiother Oncol. 2019 Mar;132:16-22. doi: 10.1016/j.radonc.2018.11.019. Epub 2018 Dec 20. PMID 30825964
- [Background] El-Bared N, Portelance L, Spieler BO, Kwon D, Padgett KR, Brown KM, Mellon EA. Dosimetric Benefits and Practical Pitfalls of Daily Online Adaptive MRI-Guided Stereotactic Radiation Therapy for Pancreatic Cancer. Pract Radiat Oncol. 2019 Jan;9(1):e46-e54. doi: 10.1016/j.prro.2018.08.010. Epub 2018 Aug 25. PMID 30149192
- [Background] Luterstein E, Cao M, Lamb J, Raldow AC, Low DA, Steinberg ML, Lee P. Stereotactic MRI-guided Adaptive Radiation Therapy (SMART) for Locally Advanced Pancreatic Cancer: A Promising Approach. Cureus. 2018 Mar 14;10(3):e2324. doi: 10.7759/cureus.2324. PMID 29765792
- [Background] Olberg S, Green O, Cai B, Yang D, Rodriguez V, Zhang H, Kim JS, Parikh PJ, Mutic S, Park JC. Optimization of treatment planning workflow and tumor coverage during daily adaptive magnetic resonance image guided radiation therapy (MR-IGRT) of pancreatic cancer. Radiat Oncol. 2018 Mar 24;13(1):51. doi: 10.1186/s13014-018-1000-7. PMID 29573744
- [Background] Tyran M, Jiang N, Cao M, Raldow A, Lamb JM, Low D, Luterstein E, Steinberg ML, Lee P. Retrospective evaluation of decision-making for pancreatic stereotactic MR-guided adaptive radiotherapy. Radiother Oncol. 2018 Nov;129(2):319-325. doi: 10.1016/j.radonc.2018.08.009. Epub 2018 Aug 30. PMID 30174107
- [Background] Rudra S, Jiang N, Rosenberg SA, Olsen JR, Roach MC, Wan L, Portelance L, Mellon EA, Bruynzeel A, Lagerwaard F, Bassetti MF, Parikh PJ, Lee PP. Using adaptive magnetic resonance image-guided radiation therapy for treatment of inoperable pancreatic cancer. Cancer Med. 2019 May;8(5):2123-2132. doi: 10.1002/cam4.2100. Epub 2019 Apr 1. PMID 30932367